CLINICAL TRIAL: NCT00228150
Title: A Phase II, Randomized, Multicenter, Double-Blind, Placebo-Controlled, Efficacy, Safety and Tolerability Study of SR57667B in Outpatients With Early Parkinson's Disease
Brief Title: Study of the Effect of SR57667B on the Progression of Symptoms in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC5287
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; levodopa; dopamine agonists
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: SR57667B

SUMMARY:
The primary objective is to assess the effect of SR57667B at the dose of 4 mg/d on the progression of Parkinson symptoms in patients with early PD. The primary outcome will be the time to progression of disability warranting initiation of L-dopa or a dopamine agonist. Secondary outcomes will comprise assessments of symptoms, activities of daily living and global clinical status.

DETAILED DESCRIPTION:
Multinational, multicenter, randomized, parallel-group, double-blind, phase II study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients.
* Age >=35 years at screening.·
* Diagnosis of Parkinson's syndrome, on at least two of the three key Parkinson's symptoms, i.e. resting tremor, bradykinesia and rigidity.
* Duration of the disease of less than 3 years since diagnosis·
* Modified Hoehn and Yahr stage <= 2.5.
* Untreated patients.
* Generally healthy and ambulatory.
* Patient has given his informed written consent and is capable of following study procedures.

Exclusion Criteria:

* Any indication of forms of parkinsonism other than PD.
* Severe resting tremor.
* Presence of either dyskinesia, fluctuations, or loss of postural reflexes·
* Treatment with L-Dopa, dopamine agonist, amantadine, anticholinergics, catechol-o-methyltransferase (COMT ) inhibitors, selegiline, dopamine receptor antagonists, catecholamine depleters, indirect dopamine agonists or alphamethyldopa.
* Electroconvulsive therapy (ECT).
* Use of CYP3A4 strong, and moderate inducers or inhibitors.
* Participation in another clinical trial with an investigational drug within two months prior to randomization.
* Dementia, uncontrolled depression, psychotic disorder.
* History of substance-related disorders including alcohol or other substance use disorders.
* Females of child bearing potential.
* Evidence (detected by history, physical examination and/or laboratory/ECG tests) of any clinically significant or unstable medical disorder that could interfere with the patient's participation in the clinical trial; interfere with the absorption, metabolism or excretion of the study medication; or interfere with the evaluation of the study drug.
* Alterations of laboratory tests or ECG findings of potential clinical significance.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2003-07; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Time to disability warranting introduction of Ldopaor a dopamine agonist.

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS)

CONTACTS AND LOCATIONS:
Overall Officials: Mark GUTMAN, MD, Study Chair — Scientific Advisory Committee; Werner POEWE, MD, Study Chair — Scientific Advisory Committee; Olivier RASCOL, MD, Study Chair — Scientific Advisory Committee; Eduardo TOLOSA, MD, Study Chair — Scientific Advisory Committee
Locations (13):
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Casablanca, Morocco
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Mégrine, Tunisia
- Sanofi-Aventis Administrative Office, Guilford Surrey, United Kingdom

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com